CLINICAL TRIAL: NCT02459171
Title: Household Transmission of Zoonotic Influenza Viruses in a Cohort of Egyptian Poultry Growers
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Human Link (Unknown)
Responsible Party: Sponsor
Other Study IDs: EGYFLU2; HHSN272201400006C (Other Grant/Funding Number: Department of Health and Human Services)
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2024-04-03 (Actual); Status verified 2023-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Surveys and Questionnaires; Blood Specimen Collection; Phlebotomy; Nasal Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects who agree to participate in this study will have blood samples collected for influenza testing, antibody determination and viral typing. Subjects will be asked for permission to keep any remaining samples for possible use in future research studies such as testing for antibodies or evidence of infection with another influenza virus or other pathogen. Some samples will be stored indefinitely at the laboratory at the National Research Centre (NRC), Egypt, or St. Jude Children's Research Hospital (SJCRH).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Subjects who meet eligibility requirements and consent to participate.
  Interventions: Blood sample, nasal wash, throat swab, questionnaire
  Interventions: Other: Questionnaire; Other: Blood sample; Other: Nasal wash; Other: Throat swab

INTERVENTIONS:
Other: Questionnaire — Once at enrollment, subjects will complete an enrollment question to capture poultry exposure and other demographic information. Information will be updated if needed at annual follow-up and at final visits.
  Other Names: Demographic information
Other: Blood sample — Participants will have a 3-mo blood sample drawn for serological testing at enrollment, and at annual follow-up and final visits.
  For subjects who test positive for influenza A by rapid test or PCR (index case) on nasal swab at the biweekly or weekly visits, two 3-ml blood samples will be obtained from the index case on day 1 for serological testing for antibodies against avian influenza viruses and for isolating and studying PBMCs. Blood samples will also be obtained on day 1 from all household contacts of the index case. Additional 3-ml blood samples will be obtained on day 14 for serology and PBMCs.
  Other Names: Blood draw; Phlebotomy
Other: Nasal wash — Nasal washes will be obtained from subjects who test positive for influenza A by rapid test or PCR on nasal swab (index case). Nasal washes will also be obtained from all household contacts of the index case. The index case and household contacts will be re-sampled on days 3, 6, 9 and 14 post initial diagnosis date.
Other: Throat swab — Throat swabs will be obtained from subjects who test positive for influenza A by rapid test or PCR on nasal swab (index case). Throat swabs will also be obtained from all household contacts of the index case. The index case and household contacts will be re-sampled on days 3, 6, 9 and 14 post initial diagnosis date.

SUMMARY:
This study seeks to determine the incidence and transmission of avian influenza viruses in humans exposed to poultry. Enrolled subjects will be selected from five different rural areas (villages) in the Nile delta region in Egypt where poultry are commonly raised. From those study sites, 2400 healthy subjects will be monitored for 6 years with annual follow up visits to measure sero-prevalence and exposure variables, and more importantly, biweekly or weekly visits to measure incidence of infection, measure secondary transmission rates, monitor symptoms, and assess immunological response.

Primary Objectives:

* To estimate the incidence of avian influenza (AI) in poultry-exposed human populations.
* To estimate sero-prevalent of AI in poultry-exposed human populations.
* To investigate potential risk factors associated with AI human infections in poultry-exposed individuals.
* To investigate secondary infection risk for household contacts.

Secondary Objectives:

* To characterize the antigenic and genetic makeup of AI viruses infecting humans.
* To monitor the pathogenicity and disease severity of AI viruses causing human infections and the associated immune response.
* To investigate the serologic response following confirmed influenza virus infection.

DETAILED DESCRIPTION:
All residents of a household will be invited to participate. After study enrollment, participants will complete a questionnaire to collect data on the demographics and health status of the subjects and the poultry kept at the household. A 3-ml blood sample will be obtained from each subject for serological testing.

Field nurses or physicians will visit each household biweekly (October through March) or weekly (April through September) to determine if any subject has influenza-like illness (ILI), defined according to Centers for Disease Control (CDC) criteria as having measured fever of ≥38ºC. and cough and/or sore throat. Subjects with confirmed ILI (index case) will provide two nasal swabs for a point-of-care rapid influenza A test and PCR. For those who test positive for influenza A by rapid test or PCR on nasal swab (day 1), two 3-ml blood samples will be obtained. In addition, nasal washes, throat swabs, and blood samples will be obtained from all household contacts.

Cloacal swabs will also be collected from the poultry in the household on day 1.

The index case and household contacts will be re-sampled by nasal wash and throat swab on days 3, 6, 9 and 14 post initial diagnosis data, and an additional 3-ml blood sample will be obtained on day 14 for serological testing.

Household contacts who report ILI symptoms during follow-up visits to the index case will then be followed with the same follow-up regimen as the original index case.

At annual follow-up and final visits, questionnaire data will be updated if needed, and a 3-ml blood sample will be obtained from each subject for serological testing.

ELIGIBILITY:
Inclusion Criteria:

* Poultry-exposed individuals with poultry in the household willing to participate by signing a consent or assent form as appropriate for age, completing the study questionnaire, and permitting the withdrawal of blood, nasal washes, nasal swabs, and throat swabs.

Exclusion Criteria:

* Any known immunosuppressive condition or immune deficiency disease (including HIV infection), or ongoing receipt of any immunosuppressive therapy. (Note that we have chosen to exclude such populations because of their increased risk of acquiring infections, they are relatively few, and are not representative of a national sample.)
* Terminally ill individuals.
* Children who are less than 2 years old when baseline enrollment is performed.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted on rural Egyptian poultry growers in areas where avian influenza is endemic in Egypt. The study sample is expected to have the same composition as the general population in that area.
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
Incidence of avian influenza (AI) in poultry-exposed populations | Up to 6 years
  New cases of avian influenza (AI) in poultry-exposed human populations will be detected using throat and nasal swabs and nasal washes obtained from subjects using rapid tests and molecular techniques.
Sero-prevalence rates of infection with AI viruses | Up to 6 years
  Prevalence rates will be measured by the presence of antibodies against AI viruses subtypes using a micro-neutralization assay. Incidence rates will be assessed based on molecular detection of AI infection annually with 95% confidence intervals. Risk or protective factors correlated with infection will be measured using the baseline enrollment questionnaire.
Risk factors associated with AI human infections in poultry-exposed individuals | Up to 6 years
  A questionnaire will be used to collect specific occupational, environmental, and behavioral risk factors. These will be correlated to sero-prevalence and incidence of AI infections.
Secondary infection risk for household contacts | Up to 6 years
  Throat and nasal swabs, blood, and nasal washes will be obtained from household contacts of poultry-exposed individuals with a confirmed influenza A infection. These will be tested for the presence of influenza A viruses or antibodies against influenza A viruses.

SECONDARY OUTCOMES:
Antigenic and genetic makeup of AI viruses infecting humans | Up to 6 years
  PCR, sequencing, culture and serological techniques will be used to characterize these viruses.
Pathogenicity and disease severity of AI viruses causing human infections and the associated immune response | Up to 6 years
  Data will be collected on disease pathogenicity and severity of symptoms from subjects reporting ILI and blood samples will be obtained to isolate and study peripheral blood mononuclear cells (PBMCs). PBMCs will be used to study innate and adaptive cell phenotyping by flow cytometry and functional assays that will be read out by flow cytometry and ELISPOT.
Serologic response following confirmed influenza virus infection | Up to 6 years
  Antibodies will be measured in acute and convalescent sera of confirmed influenza cases.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Webby, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- National Research Centre, Cairo, Egypt

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols